CLINICAL TRIAL: NCT03805386
Title: Patient-Directed Postoperative Opioid Prescribing for Gynecologic Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Johnny Yi, Prinicpal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-004216
Record Dates: First submitted 2019-01-12; First posted 2019-01-15 (Actual); Results first posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-01

CONDITIONS: Gynecology; Surgery; Opioid Use
Keywords: patient directed postoperative opioid prescribing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (Active Comparator): Subjects will be prescribed the standard amount of opioids that are typically prescribed by our practice after surgery. Oxycodone 5mg 1-2 tablets every 4 hours as needed for pain. 30 tablets will be provided.
  Interventions: Drug: Physician directed opioid prescribing
- Patient Directed Care (Experimental): Subject directed arm will be prescribed the number of opioids that the patient decides to be appropriate after discussion with the surgeon. This can be as low as 0 pills and as much as 30 pills as described in the standard care.
  Interventions: Drug: Patient directed opioid prescribing

INTERVENTIONS:
Drug: Physician directed opioid prescribing — Oxycodone 5mg 1-2 tablets every 4 hours as needed for pain. 30 tablets will be provided.
  Arms: Standard of Care
Drug: Patient directed opioid prescribing — Oxycodone 5mg amount ranging from 0 tablets to as much as 30 tablets as described in the standard of care.
  Arms: Patient Directed Care

SUMMARY:
We would like to evaluate and optimize opioid prescribing after minimally invasive hysterectomy. Currently, our standard prescribing is 150 oral morphine equivalents. However, recent studies show that half of the opioids prescribed are not used. We would like to include the patient in the decision making of the opioid prescribing.

We have designed a randomized controlled trial to prescribe standard (150 oral morphine equivalents) or patient directed (less than or equal to 150 oral morphine equivalents) for pain control.

We hypothesize that with patient input, there will be a higher utilization of the opioids prescribed. Also, we anticipate a lower number of opioids used overall.

This study will help us optimize opioid prescribe and evaluate whether patient input can help in this important measure.

DETAILED DESCRIPTION:
There is an emphasis in patient centered care in medicine and part of this effort has evaluated the success of shared decision making in the care of the patient. Currently, there is strong research and clinical emphasis trying to determine how, as surgeons, we can assist in minimizing the misuse of opioid medications. Several studies have shown significant over-prescribing and under-utilizing of the pain medications that are prescribed to patients after surgery. One such study by As-Sanie et al showed that about half of medications were utilized for pain after surgery, with typically 200 oral morphine equivalents prescribed.

A recent prospective cohort study by Prabhu et al showed that shared decision making in the prescription of narcotic pain medications after cesarean section decreased opioid use without impacting patient satisfaction.

We propose a randomized controlled trial evaluating the impact of shared decision making in the prescribing of pain medications after minimally invasive gynecologic surgery. For adult female patients who are undergoing minimally invasive hysterectomy, we will randomize them to either standard care or patient directed treatment. Our standard arm will receive 150 oral morphine equivalents, or 30 tablets of oxycodone, whereas our patient directed arm will receive a prescription with as many pills is determined after discussion with the patient.

We hope to contribute to identifying the optimized opioid prescription for post surgical patients.

ELIGIBILITY:
Inclusion criteria

* Female patients >18 years old
* Ability to provide informed consent
* Planned minimally invasive hysterectomy with the Department of Gynecology o Concomitant minimally invasive surgeries performed by Gynecology will be allowed

Exclusion criteria

* Non-English speaking
* Combined surgical cases with other surgical departments
* Planned laparotomy
* Surgery planned to last >4 hours
* Postoperative hospitalization planned for >7 days
* Planned use of oral opioids other than oxycodone postoperatively
* Pre-existing chronic pain conditions including: chronic pelvic pain, migraines, temporomandibular joint dysfunction syndrome, fibromyalgia, and interstitial cystitis
* Preoperative diagnosis of pelvic pain
* Chronic preoperative opioid use
* History of or current diagnosis of narcotic or alcohol dependence

  o Screening question asked at preoperative appointment: Have you or are you currently dependent on narcotic medications or alcohol?
* Desire for more opioids than standard therapy
* Postoperative decision of surgeon to prescribed more than standard therapy
* Allergy or contraindication to taking opioids, ibuprofen, or acetaminophen

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnny Yi, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ambulatory Gynecologic Surgery Clinic
Groups:
- Patient Directed Care: Subject directed arm will be prescribed the number of opioids that the patient decides based on shared decision making model to be appropriate after discussion with the surgeon. This can be as low as 0 pills and as much as 30 pills as described in the standard care.
  Patient directed opioid prescribing: Oxycodone 5mg amount ranging from 0 tablets to as much as 30 tablets as described in the standard of care.
Period: Overall Study
Arm/Group | Standard of Care | Patient Directed Care
Started | 32 | 33
Completed | 32 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Patient Directed Care: Subject directed arm will be prescribed the number of opioids that the patient decides based on a shared decision making model to be appropriate after discussion with the surgeon. This can be as low as 0 pills and as much as 30 pills as described in the standard care.
  Patient directed opioid prescribing: Oxycodone 5mg amount ranging from 0 tablets to as much as 30 tablets as described in the standard of care.
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Patient Directed Care | Total
Number analyzed (Participants) | 32 | 33 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 24 | 44
  >=65 years | 12 | 9 | 21
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59.5 [50 to 66.5] | 52 [46 to 64] | 55 [47 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 33 | 65
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | NA — Did not ask | NA — did not ask | NA — Total not calculated because data are not available (NA) in one or more arms.
  Black or African American | 0 | 2 | 2
  White | 28 | 29 | 57
  More than one race | NA — did not ask | NA — did not ask | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 32 | 33 | 65
BMI [Median (Inter-Quartile Range); unit: kg/m2] | 26.3 [24 to 33.1] | 28.3 [24.5 to 33.1] | 26.9 [24 to 33.1]

OUTCOME MEASURES:

1. Primary Outcome: # of Opioid Pills Consumed
Description: Percent utilization of opioids consumed (consumed/prescribed)
Time Frame: 6 weeks postop
Measure: Mean (Standard Error); unit: % oxycodone used
Arm/Group | Standard of Care | Patient Directed Care
Number analyzed (Participants) | 32 | 33
% oxycodone used | 26.7 (0.91) | 38.4 (1.08)

2. Secondary Outcome: Opioid Pills Prescribed
Description: Number of opioids prescribed
Time Frame: preoperative visit
Measure: Median (Inter-Quartile Range); unit: pills
Groups:
- # Pills Prescribed Standard: The number of 5mg oxycodone pills prescribed to patients at the preoperative visit.
- # Pills Prescribed Patient Directed: # of 5mg oxycodone pills prescribed based on shared decision making.
Arm/Group | # Pills Prescribed Standard | # Pills Prescribed Patient Directed
Number analyzed (Participants) | 32 | 33
pills | 30 [30 to 30] | 15 [12 to 24]

3. Secondary Outcome: Patient Satisfaction
Description: Patients were asked if they were satisfied with the # of oxycodone pills prescribed.
Time Frame: 6 weeks post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Patient Directed Care
Number analyzed (Participants) | 32 | 33
Participants | 27 | 29

ADVERSE EVENTS:
Time Frame: Patients were followed up to 6 weeks postoperative visit.
Arm/Group | Standard of Care | Patient Directed Care
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/33
Other Adverse Events (participants affected / at risk) | 0/32 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-29): https://cdn.clinicaltrials.gov/large-docs/86/NCT03805386/Prot_SAP_000.pdf